CLINICAL TRIAL: NCT03963856
Title: MULTI-SYSTEM PHYSIOLOGIC RESPONSE TO VARYING LEVELS OF PARTIAL GRAVITY
Acronym: GRAVIDOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-072
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: parbolic flight — weightlessness during parabolic flight

SUMMARY:
Spaceflight induces detrimental changes in most organ systems with both acute changes and chronic adaptations. For example, acute fluid shifts associated with weightlessness (also called - improperly - microgravity) cause initial rapid cardiovascular alterations, whereas the chronic changes are more reflective of cardiovascular deconditioning and cerebrovascular/ocular adaptations (Pavy-Le Traon et al., 2007).

Long-duration stays in weightlessness have resulted in ocular structural and functional adaptations in some astronauts, which has been termed the Spaceflight Associated Neuro-ocular Syndrome (SANS ; see review in Lee et al., 2018). The leading hypothesis is that ocular changes are the consequence of chronic exposure to the weightlessness-induced headward (cephalad) fluid shift experienced by all astronauts. Countermeasures targeted to reverse this fluid shift, including lower body negative pressure and veno-occlusive thigh cuffs, have been proposed and tested in ground-based studies using a head-down tilt model of the cephalad fluid shift. However, the amount of fluid shift reversal required to prevent the development of SANS has not been investigated or determined. Similarly, artificial gravity through centrifugation has been proposed as a SANS countermeasure, given its ability to reverse headward fluid shifts and its efficacy as a countermeasure to long-duration bed rest-induced cardiovascular adaptations (long-duration bed rest is widely employed to simulate the effects of microgravity on various physiological systems). However, the minimum level of artificial gravity required also has not been investigated.

The primary objective of this study is to characterize cardiovascular, cerebrovascular, and ocular changes across a range of gravity levels to identify a threshold of gravitational load that can serve as a countermeasure to SANS during future spaceflight missions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who have passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Persons who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women (urine pregnancy test for women of childbearing potential)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | baseline
  will be assessed continuously using the Triggerfish

CONTACTS AND LOCATIONS:
Locations (1):
- CHU caen, Caen, France

IPD SHARING:
Plan to Share IPD: No